CLINICAL TRIAL: NCT06033521
Title: Treatment Patterns of Menopausal Hormone Therapy in South Korea: a Nationwide Cohort Study
Brief Title: A Study to Learn More About the Menopausal Hormone Therapies in Korea
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B2311076; MHT RWD (Other: Alias Study Number)
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Menopause; Bone Demineralization
Keywords: Menopause; Bone Demineralization; Hormone Replacement Therapy
MeSH Terms: conditions — Bone Demineralization, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with menopausal hormone therapy: Subjects who were newly diagnosed menopausal symptoms between 01 Jan 2012 and 31 Dec 2019, and were followed up for 12 months at least in the HIRA claims database
  Interventions: Drug: Menopausal hormone therapy Intervention Type: Drug

INTERVENTIONS:
Drug: Menopausal hormone therapy Intervention Type: Drug — Subjects who were newly diagnosed menopausal symptoms between 01 Jan 2012 and 31 Dec 2019, and were followed up for 12 months at least in the HIRA claims database

SUMMARY:
The purpose of this study is to learn about how the commonly used menopausal hormone therapies were prescribed and taken in practice. This is done by using healthcare database, to study the overall dangers and benefits of menopausal hormone therapies in real-world practice.

This study will include subjects who were newly diagnosed menopausal symptoms between 2012 and 2019. They were all followed up for 12 months at least.

The study included the below subjects who:

* were aged 40-59 years
* were diagnosed to have menopausal symptoms through some medical check-ups

The data collected will be used to understand:

* how the commonly used menopausal hormone therapies were prescribed and taken in practice
* how patients took medication as prescribed by their doctors This might help to understand treatment trends of these therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-59 years at cohort entry date
* Patients who had at least one inpatient or outpatient diagnosis of menopausal symptoms between 01 Jan 2012 and 31 Dec 2019 with any of following diagnosis codes: N95.1, N95.2, N95.3, N95.8, N95.9, M80.0, M81.0, M81.99, M85.99

Exclusion Criteria:

* Patients diagnosed with breast cancer (C50, D05), endometrial cancer (C54.1), and granulosa cell tumor (C56) within 1 year prior to the index date.
* Patients diagnosed with coronary heart disease (I20-I25, I51.6), stroke (I60-64), and VTE (I80.2, I80.3 I26) within 1 year prior to the index date.
* Patients diagnosed with viral hepatitis (B16-B19), cirrhosis (K70.2-K70.4, K71.7, K72.0-K72.1, K72.9, K74.0-K74.6, K76.1, K76.6-K76.7, R18, I85.0, I85.9, I86.4, I86.8, I98.2-I98.3), and hepatic cancer (C22) within 1 year prior to the index date.
* Patients diagnosed with gallbladder disease (K80, K81, K82, K83, K85.1), gallbladder cancer (C23), extrahepatic bile duct cancer (C24) within 1 year prior to the index date.

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Subjects who were newly diagnosed menopausal symptoms between 01 Jan 2012 and 31 Dec 2019, and were followed up for 12 months at least in the HIRA claims database
Sampling Method: Probability Sample
Enrollment: 1036294 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer South Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B2311076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data for female participants in South Korea, aged 40-59 years who had diagnosis of menopausal symptoms and/or received menopausal hormone therapy (MHT), was retrieved from Health Insurance and Review Assessment (HIRA) database from 1-January-2016 and 31-Decemeber-2020 (included follow-up duration). Retrospective available data was evaluated as per objectives of this study from 12-September-2023 to 11-March-2024 (approximately 6 months).
Groups:
- All Participants: Female participants aged 40-59 years who had diagnosis of menopausal symptoms and/or received MHT in real-world practice. No intervention was administered during this study.
Period: Overall Study
Arm/Group | All Participants
Started | 1036294
Completed | 1036294
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants who met inclusion/exclusion criteria, whose data were included and observed for evaluation in the study.
Groups:
- Participants With MHT: Female participants aged 40-59 years who had diagnosis of menopausal symptoms and received MHT in real-world practice. No intervention was administered during this study.
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.53 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1036294
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Who Visited Hospitals for Menopausal Symptoms Distributed Per Year
Description: Menopausal symptoms: at least one inpatient or outpatient claim with any of diagnosis codes based on Korean standard classification of disease, 8th revision(KCD-8):Korean version of ICD-10(International statistical classification of diseases and related health problems,10th revision), per protocol. N95.1: Menopausal, female climacteric states; N95.2:Postmenopausal atrophic vaginitis; N95.3:States associated with artificial menopause; N95.8 Other specified menopausal, perimenopausal disorders; N95.9: Menopausal, perimenopausal disorder, unspecified; M80.0: Postmenopausal osteoporosis with pathological fracture;M81.0: Postmenopausal osteoporosis; M81.99:Osteoporosis, unspecified, site unspecified; Osteopenia; M85.99: Disorder of bone density, structure, unspecified, site unspecified; Osteopenia, mild; Osteopenia, moderate; Osteopenia, severe. One participant could have visited hospital for >=1 time for different menopausal symptom. Index date: date of first prescription for MHT.
Time Frame: Date of diagnosis of menopausal symptom during inpatient/outpatient hospital visit; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Participants
  2016 | 786616
  2017 | 787425
  2018 | 791890
  2019 | 818749

2. Primary Outcome: Number of Women With MHT Use Distributed Per Year
Description: Number of Women with MHT use distributed per year was reported in this outcome measure. One participant could have taken more than 1 type of MHT hence participants are not fully exclusive. Three types of MHT included ET (estrogen therapy), EPT (estrogen-progestin therapy), and tibolone. Index date was defined as the date of the first prescription for MHT.
Time Frame: Index Date; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Participants
  2016 | 446702
  2017 | 473592
  2018 | 481568
  2019 | 494192

3. Primary Outcome: Number of Participants According to Each Type of Menopausal Symptoms Distributed Per Year
Description: Menopausal symptoms included vasomotor, bone and joint, genitourinary and psychosomatic. One participant could have more than 1 type of menopausal symptoms. Index date was defined as the date of the first prescription for MHT.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants who met inclusion/exclusion criteria, whose data were included and observed for evaluation in the study. Here, 'Number Analyzed' signifies participants evaluable at specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Participants
  Vasomotor: 2016: number analyzed (Participants) | 436796
  Vasomotor: 2016 | 358505
  Bone and joint: 2016: number analyzed (Participants) | 436796
  Bone and joint: 2016 | 28208
  Genitourinary: 2016: number analyzed (Participants) | 436796
  Genitourinary: 2016 | 80857
  Psychosomatic: 2016: number analyzed (Participants) | 436796
  Psychosomatic: 2016 | 1809
  Vasomotor: 2017: number analyzed (Participants) | 435597
  Vasomotor: 2017 | 119084
  Bone and joint: 2017: number analyzed (Participants) | 435597
  Bone and joint: 2017 | 8396
  Genitourinary: 2017: number analyzed (Participants) | 435597
  Genitourinary: 2017 | 57812
  Psychosomatic: 2017: number analyzed (Participants) | 435597
  Psychosomatic: 2017 | 780
  Vasomotor: 2018: number analyzed (Participants) | 424687
  Vasomotor: 2018 | 92169
  Bone and joint: 2018: number analyzed (Participants) | 424687
  Bone and joint: 2018 | 6635
  Genitourinary: 2018: number analyzed (Participants) | 424687
  Genitourinary: 2018 | 48640
  Psychosomatic: 2018: number analyzed (Participants) | 424687
  Psychosomatic: 2018 | 648
  Vasomotor: 2019: number analyzed (Participants) | 423547
  Vasomotor: 2019 | 85728
  Bone and joint: 2019: number analyzed (Participants) | 423547
  Bone and joint: 2019 | 6025
  Genitourinary: 2019: number analyzed (Participants) | 423547
  Genitourinary: 2019 | 42798
  Psychosomatic: 2019: number analyzed (Participants) | 423547
  Psychosomatic: 2019 | 652

4. Primary Outcome: Number of Participants According to Each Type of Menopausal Symptoms Per MHT
Description: Menopausal symptoms included vasomotor symptoms, bone and joint symptoms, genitourinary symptoms, psychosomatic symptoms for systemic, Estrogen Therapy (ET), Estrogen-Progestin Therapy (EPT) and Tibolone. One participant could have more than 1 type of menopausal symptoms and have received more than 1 type of therapy. Index date was defined as the date of the first prescription for MHT.
Time Frame: Index Date; retrospective data observed in this study for approximately 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Participants
  Systemic MHT: Vasomotor symptoms: number analyzed (Participants) | 695824
  Systemic MHT: Vasomotor symptoms | 649307
  Systemic MHT: Bone and joint symptoms: number analyzed (Participants) | 695824
  Systemic MHT: Bone and joint symptoms | 83856
  Systemic MHT: Genitourinary symptoms: number analyzed (Participants) | 695824
  Systemic MHT: Genitourinary symptoms | 44385
  Systemic MHT: Psychosomatic symptoms: number analyzed (Participants) | 695824
  Systemic MHT: Psychosomatic symptoms | 4951
  ET: Vasomotor symptoms: number analyzed (Participants) | 89237
  ET: Vasomotor symptoms | 80044
  ET: Bone and joint symptoms: number analyzed (Participants) | 89237
  ET: Bone and joint symptoms | 12479
  ET: Genitourinary symptoms: number analyzed (Participants) | 89237
  ET: Genitourinary symptoms | 8087
  ET: Psychosomatic symptoms: number analyzed (Participants) | 89237
  ET: Psychosomatic symptoms | 710
  EPT: Vasomotor symptoms: number analyzed (Participants) | 300999
  EPT: Vasomotor symptoms | 287092
  EPT: Bone and joint symptoms: number analyzed (Participants) | 300999
  EPT: Bone and joint symptoms | 30659
  EPT: Genitourinary symptoms: number analyzed (Participants) | 300999
  EPT: Genitourinary symptoms | 16825
  EPT: Psychosomatic symptoms: number analyzed (Participants) | 300999
  EPT: Psychosomatic symptoms | 2241
  Tibolone: Vasomotor symptoms: number analyzed (Participants) | 306538
  Tibolone: Vasomotor symptoms | 283069
  Tibolone: Bone and joint symptoms: number analyzed (Participants) | 306538
  Tibolone: Bone and joint symptoms | 40833
  Tibolone: Genitourinary symptoms: number analyzed (Participants) | 306538
  Tibolone: Genitourinary symptoms | 19581
  Tibolone: Psychosomatic symptoms: number analyzed (Participants) | 306538
  Tibolone: Psychosomatic symptoms | 2021

5. Primary Outcome: Number of Participants With Use of Any MHT According to Age Group
Description: Number of participants with use of any MHT according to age group were reported in this outcome measure. Index date was defined as the date of the first prescription for MHT.
Time Frame: Index Date; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Participants
  40-44 Years | 39917
  45-49 Years | 199389
  50-54 Years | 425030
  55-59 Years | 371958

6. Primary Outcome: Number of Participants With MHT According to Type of Administration
Description: Number of participants with MHT according to type of administration were reported in this outcome measure. Type of administration included systemic hormone therapy (HT) (oral), systemic HT (transdermal), local HT (transvaginal). One participant could have received more than 1 type of therapy. Index date was defined as the date of the first prescription for MHT.
Time Frame: Index Date; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Participants
  Systemic MHT (oral) | 693072
  Systemic MHT (transdermal) | 2960
  Local MHT (transvaginal) | 378764

7. Primary Outcome: Percentage of Participants With Change in Treatment Regimen Change at Month 3
Description: Percentage of participants with change in treatment regimen at Month 3 were reported in this outcome measure. Data reported in this outcome measure included participants who received the treatments which included Systemic ET, EPT, Tibolone, Local ET and also participants with no treatment. Index date was defined as the date of the first prescription for MHT.
Time Frame: Month 3 post-index date; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic ET | 5.8
  EPT | 17.6
  Tibolone | 20.4
  Local ET | 4.1
  No treatment provided | 52.1

8. Primary Outcome: Percentage of Participants With Change in Treatment Regimen Change at Month 6
Description: Percentage of participants with change in treatment regimen at Month 6 were reported in this outcome measure. Data reported in this outcome measure included participants who received the treatments which included Systemic ET, EPT, Tibolone, Local ET and also participants with no treatment. Index date was defined as the date of the first prescription for MHT.
Time Frame: Month 6 post-index date; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic ET | 4.3
  EPT | 11.0
  Tibolone | 14.0
  Local ET | 0.9
  No treatment provided | 69.8

9. Primary Outcome: Percentage of Participants With Change in Treatment Regimen Change at Month 9
Description: Percentage of participants with change in treatment regimen at Month 9 were reported in this outcome measure. Data reported in this outcome measure included participants who received the treatments which included Systemic ET, EPT, Tibolone, Local ET and also participants with no treatment. Index date was defined as the date of the first prescription for MHT.
Time Frame: Month 9 post-index date; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic ET | 3.5
  EPT | 8.5
  Tibolone | 11.1
  Local ET | 0.6
  No treatment provided | 76.3

10. Primary Outcome: Percentage of Participants With Change in Treatment Regimen Change at Month 12
Description: Percentage of participants with change in treatment regimen at Month 12 were reported in this outcome measure. Data reported in this outcome measure included participants who received the treatments which included Systemic ET, EPT, Tibolone, Local ET and also participants with no treatment. Index date was defined as the date of the first prescription for MHT.
Time Frame: Month 12 post-index date; retrospective data observed in this study for approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic ET | 3.0
  EPT | 7.0
  Tibolone | 9.4
  Local ET | 0.5
  No treatment provided | 80.1

11. Primary Outcome: Time to Discontinuation of MHT
Description: Time to discontinuation was defined as no subsequent prescriptions within 2 months of last prescription date. MHT included: Systemic MHT: ET, EPT, Tibolone and Local MHT: ET. Index date was defined as the date of the first prescription for MHT.
Time Frame: During 2 year of follow up from index date; retrospective data observed in this study for approximately 6 months
Population: Analysis population included all eligible participants who met inclusion/exclusion criteria, whose data were included and observed for evaluation in the study. Here, 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Months
  Systemic MHT: ET: number analyzed (Participants) | 89237
  Systemic MHT: ET | 14.4 (17.7)
  Systemic MHT: EPT: number analyzed (Participants) | 300999
  Systemic MHT: EPT | 10.1 (13.7)
  Systemic MHT: Tibolone: number analyzed (Participants) | 306538
  Systemic MHT: Tibolone | 13.4 (16.6)
  Local MHT: ET: number analyzed (Participants) | 378764
  Local MHT: ET | 2.4 (1.2)

12. Primary Outcome: Time to Switching of MHT
Description: Time to switching of MHT was reported in this outcome measure. Participants who switched the treatment classes were included. MHT included: Systemic MHT: ET, EPT, Tibolone and Local MHT: ET. Index date was defined as the date of the first prescription for MHT.
Time Frame: During 2 year of follow up from index date; retrospective data observed in this study for approximately 6 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Months
  Systemic MHT: ET: number analyzed (Participants) | 89237
  Systemic MHT: ET | 13.2 (15.0)
  Systemic MHT: EPT: number analyzed (Participants) | 300999
  Systemic MHT: EPT | 16.9 (15.5)
  Systemic MHT: Tibolone: number analyzed (Participants) | 306538
  Systemic MHT: Tibolone | 13.9 (14.7)
  Local MHT: ET: number analyzed (Participants) | 378764
  Local MHT: ET | 7.1 (11.7)

13. Primary Outcome: Percentage of Participants With Treatment Persistence at Month 3 Post-index According to Treatment Type
Description: Treatment persistence was calculated by the average length of treatment of the drugs prescribed at the index date. Index date was defined as the date of the first prescription for MHT.
Time Frame: Month 3 post-index; retrospective data observed in this study for approximately 6 months
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic MHT: ET: number analyzed (Participants) | 89237
  Systemic MHT: ET | 69.5 [upper limit 22.1]
  Systemic MHT: EPT: number analyzed (Participants) | 300999
  Systemic MHT: EPT | 60.9 [3.2 to 27.7]
  Systemic MHT: Tibolone: number analyzed (Participants) | 306538
  Systemic MHT: Tibolone | 75.8 [1.2 to 22.5]
  Local MHT: ET: number analyzed (Participants) | 378764
  Local MHT: ET | 11.8 [0.0 to 10.6]

14. Primary Outcome: Percentage of Participants With Treatment Persistence at Month 6 Post-index According to Treatment Type
Description: as for outcome 13
Time Frame: Month 6 post-index; retrospective data observed in this study for approximately 6 months
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic MHT: ET: number analyzed (Participants) | 89237
  Systemic MHT: ET | 48.2 [upper limit 22.1]
  Systemic MHT: EPT: number analyzed (Participants) | 300999
  Systemic MHT: EPT | 36.7 [3.2 to 27.7]
  Systemic MHT: Tibolone: number analyzed (Participants) | 306538
  Systemic MHT: Tibolone | 46.4 [1.2 to 22.5]
  Local MHT: ET: number analyzed (Participants) | 378764
  Local MHT: ET | 1.1 [0.0 to 10.6]

15. Primary Outcome: Percentage of Participants With Treatment Persistence at Month 9 Post-index According to Treatment Type
Description: as for outcome 13
Time Frame: Month 9 post-index; retrospective data observed in this study for approximately 6 months
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic MHT: ET: number analyzed (Participants) | 89237
  Systemic MHT: ET | 38.7 [upper limit 22.1]
  Systemic MHT: EPT: number analyzed (Participants) | 300999
  Systemic MHT: EPT | 27.9 [3.2 to 27.7]
  Systemic MHT: Tibolone: number analyzed (Participants) | 306538
  Systemic MHT: Tibolone | 36.4 [1.2 to 22.5]
  Local MHT: ET: number analyzed (Participants) | 378764
  Local MHT: ET | 0.4 [0.0 to 10.6]

16. Primary Outcome: Percentage of Participants With Treatment Persistence at Month 12 Post-index According to Treatment Type
Description: as for outcome 13
Time Frame: Month 12 post-index; retrospective data observed in this study for approximately 6 months
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of participants
  Systemic MHT: ET: number analyzed (Participants) | 89237
  Systemic MHT: ET | 33.1 [upper limit 22.1]
  Systemic MHT: EPT: number analyzed (Participants) | 300999
  Systemic MHT: EPT | 22.6 [3.2 to 27.7]
  Systemic MHT: Tibolone: number analyzed (Participants) | 306538
  Systemic MHT: Tibolone | 30.3 [1.2 to 22.5]
  Local MHT: ET: number analyzed (Participants) | 378764
  Local MHT: ET | 0.2 [0.0 to 10.6]

17. Primary Outcome: Mean Treatment Adherence (%)
Description: Treatment adherence was evaluated using medication possession ratio (MPR), calculated as the total number of days of medication supply divided by the number of days in the follow-up period. Data for this outcome is expressed in percentage. Index date was defined as the date of the first prescription for MHT.
Time Frame: Index Date; retrospective data observed in this study for approximately 6 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Participants With MHT
Number analyzed (Participants) | 1036294
Percentage of days
  Systemic MHT: ET: number analyzed (Participants) | 89237
  Systemic MHT: ET | 37.3 (45.5)
  Systemic MHT: EPT: number analyzed (Participants) | 300999
  Systemic MHT: EPT | 22.4 (39.0)
  Systemic MHT: Tibolone: number analyzed (Participants) | 306538
  Systemic MHT: Tibolone | 35.5 (55.0)
  Local MHT: ET: number analyzed (Participants) | 378764
  Local MHT: ET | 3.1 (27.2)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be evaluated for the study.
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (that is, identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence adverse events were not planned to be evaluated (thus at risk appears "0").
Arm/Group | Participants With MHT
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT06033521/Prot_SAP_000.pdf